CLINICAL TRIAL: NCT06059365
Title: Randomized Clinical Trial to Test the Efficacy and Safety of Outpatient Clinical Management of Urgent Laparoscopic Appendectomy in Complicated Acute Appendicitis
Brief Title: Clinical Trial for a Outpatient Clinical Management for Complicated Acute Appendicitis
Acronym: ASI2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HJ23 (Industry)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Jordi Elvira Lopez, MD PhD, HJ23
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASI-2
Record Dates: First submitted 2023-09-23; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Appendicitis; Appendicitis Perforated; Appendicitis Suppurative
MeSH Terms: conditions — Appendicitis | interventions — Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hospitalization group (Active Comparator): Patients in the hospitalization group, once the surgical intervention was finished, were transferred to the postoperative recovery unit and later they were discharged to the usual hospital ward. Patients received adequate intravenous fluid resuscitation based on their individual hemodynamic parameter and fluid balance, and they received analgesia according to personal requirement. In the hospital ward, the usual patient management protocols were followed until a complete recovery and consequently discharged according to the usual criteria
  Interventions: Behavioral: Hospitalization
- outpatient group (Experimental): Patients in the outpatient group , once operated, were transferred to the surgery unit without admission and were later discharged home if they met the ALDRETE criteria in less than 23 hours after the intervention (following the surgery criteria without admission stages). If the patient was operated during the night shift, following the advice of major outpatient surgery where overnight stays are allowed, the patient was admitted to the post-anesthetic recovery unit and discharged the next day, always in less than 23 hours. In case of being discharged after 23 hours or not meeting ALDRETE criteria, it was considered a failure of the outpatient treatment.
  Interventions: Behavioral: Outpatient

INTERVENTIONS:
Behavioral: Hospitalization — Once the patient was operated and an uncomplicated appendicitis was confirmed, the patient was randomized to one of the two experimental branches: the hospitalization group (HG) or outpatient group (OG). In this group, were admitted in the hospitalization ward
  Arms: hospitalization group
Behavioral: Outpatient — Once the patient was operated and an uncomplicated appendicitis was confirmed, the patient was randomized to one of the two experimental branches: the hospitalization group (HG) or outpatient group (OG). Patients in the OG were referred to the day- surgery unit where they were discharged according to ALDRETE criteria.
  Arms: outpatient group

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of outpatient management of complicated acute appendicitis. For this purpose, a randomized clinical trial was designed. Selected patients who have undergone surgery for acute appendicitis are randomized into two groups. One group with hospitalization and another group without admission.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy and safety of outpatient management of laparoscopic appendicectomy in complicated acute appendicitis.

This was a single center randomized controlled clinical trial consisting in 2 treatment groups. Patients were recruited in University Hospital of Tarragona Joan XXIII of Spain.

All patients admitted in the emergency department at University Hospital of Tarragona Joan XXIII with acute appendicitis diagnosis were likely to enter in the study.

All patients who met the inclusion criteria and none of the exclusion criteria were admitted to the study for emergency surgery.

In order to avoid the biases a unique anesthetic and surgical protocol were established for both groups.

Once Laparoscopic appendicectomy was performed the patients were randomly assigned to the hospitalization group or outpatient group.

Patients in the hospitalization group were admitted in the hospitalization ward. Patients in the outpatient group were referred to the day-surgery unit where they were discharged according to ALDRETE criteria.

The primary endpoint was the length of hospital stay (LHS). The length of hospital stay was calculated from the day and hour of admission in the surgical area to the day and hour of discharge, based on the hours of hospital stay. Secondary endpoints included the failures of the outpatient management, readmissions and the hospitals cost

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* ASA classification (American Society of Anesthesiologists) less than or equal to 3
* patients who live accompanied in a home at a maximum distance of 30 minutes from the hospital and an adequate cognitive capacity.

Exclusion Criteria:

* pregnancy or breastfeeding
* complicated Acute Appendicitis
* surgical management performed in more 90 minutes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients over 18 years old
Enrollment: 92 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
length of hospital stay (LHS) | up to 5 days
  The length of hospital stay (LHS) was calculated from the date and time of urgent appendectomy surgery to the date and time of hospital discharge, based on the hours of hospital stay (assessed up to 5 days)

SECONDARY OUTCOMES:
failures of the outpatient management | assessed up to 30 days
  Once the patients were discharged home, they were evaluated for emergency room visit. From the date of hospital discharge to the day of emergency room visit. The presence of a emergency room visit is considered as a Failure of the outpatient management.
readmissions | assessed up to 30 days
  Once the patients were discharged home, they were evaluated for readmission to the hospital ward. From the date of hospital discharge to the day of readmission to the hospital ward. The re-admission to the hospitalization ward was considered a readmission.
hospitals cost | through study completion, an average of 1 year
  The economic costs of both clinical managements were evaluated until the end of the study, a mean of 1 year. For the study, the direct and indirect costs of laparoscopic surgery, consumable material, economic expenses in the hospital ward, and the cost of the price of the emergency room visit were evaluated. The hospital's economic department was contacted and they calculated the cost in euros per patient. Each group was evaluated separately and a comparison was made

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Elvira Lopez, MD, PhD, Principal Investigator — HJ23

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lefrancois M, Lefevre JH, Chafai N, Pitel S, Kerger L, Agostini J, Canard G, Tiret E. Management of Acute Appendicitis in Ambulatory Surgery: Is It Possible? How to Select Patients? Ann Surg. 2015 Jun;261(6):1167-72. doi: 10.1097/SLA.0000000000000795. PMID 24950287
- [Background] Frazee RC, Roberts JW, Symmonds RE, Snyder SK, Hendricks JC, Smith RW, Custer MD 3rd, Harrison JB. A prospective randomized trial comparing open versus laparoscopic appendectomy. Ann Surg. 1994 Jun;219(6):725-8; discussion 728-31. doi: 10.1097/00000658-199406000-00017. PMID 8203983
- [Background] Cash CL, Frazee RC, Smith RW, Davis ML, Hendricks JC, Childs EW, Abernathy SW. Outpatient laparoscopic appendectomy for acute appendicitis. Am Surg. 2012 Feb;78(2):213-5. PMID 22369831
- [Background] Aubry A, Saget A, Manceau G, Faron M, Wagner M, Tresallet C, Riou B, Lucidarme O, le Sache F, Karoui M. Outpatient Appendectomy in an Emergency Outpatient Surgery Unit 24 h a Day: An Intention-to-Treat Analysis of 194 Patients. World J Surg. 2017 Oct;41(10):2471-2479. doi: 10.1007/s00268-017-4034-3. PMID 28474273
- [Background] Di Saverio S, Podda M, De Simone B, Ceresoli M, Augustin G, Gori A, Boermeester M, Sartelli M, Coccolini F, Tarasconi A, De' Angelis N, Weber DG, Tolonen M, Birindelli A, Biffl W, Moore EE, Kelly M, Soreide K, Kashuk J, Ten Broek R, Gomes CA, Sugrue M, Davies RJ, Damaskos D, Leppaniemi A, Kirkpatrick A, Peitzman AB, Fraga GP, Maier RV, Coimbra R, Chiarugi M, Sganga G, Pisanu A, De' Angelis GL, Tan E, Van Goor H, Pata F, Di Carlo I, Chiara O, Litvin A, Campanile FC, Sakakushev B, Tomadze G, Demetrashvili Z, Latifi R, Abu-Zidan F, Romeo O, Segovia-Lohse H, Baiocchi G, Costa D, Rizoli S, Balogh ZJ, Bendinelli C, Scalea T, Ivatury R, Velmahos G, Andersson R, Kluger Y, Ansaloni L, Catena F. Diagnosis and treatment of acute appendicitis: 2020 update of the WSES Jerusalem guidelines. World J Emerg Surg. 2020 Apr 15;15(1):27. doi: 10.1186/s13017-020-00306-3. PMID 32295644
- [Background] Trejo-Avila M, Cardenas-Lailson E, Valenzuela-Salazar C, Herrera-Esquivel J, Moreno-Portillo M. Ambulatory versus conventional laparoscopic appendectomy: a systematic review and meta-analysis. Int J Colorectal Dis. 2019 Aug;34(8):1359-1368. doi: 10.1007/s00384-019-03341-y. Epub 2019 Jul 5. PMID 31273450
- [Background] Elvira Lopez J, Sales Mallafre R, Padilla Zegarra E, Carrillo Luna L, Ferreres Serafini J, Tully R, Memba Ikuga R, Jorba Martin R. Outpatient management of acute uncomplicated appendicitis after laparoscopic appendectomy: a randomized controlled trial. World J Emerg Surg. 2022 Nov 23;17(1):59. doi: 10.1186/s13017-022-00465-5. PMID 36419071